CLINICAL TRIAL: NCT06387173
Title: Registry of Patients Undergoing Cryoablation for Early Stage Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-001743; NCI-2024-01240 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-03-25; First posted 2024-04-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Early Stage Breast Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the side effects and outcomes of patients who undergo cryoablation for early stage breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To obtain observational real-life data of patients who choose this non-conventional treatment and to follow their outcomes.

OUTLINE: This is an observational study.

Patients have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cryoablation for breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cryoablation for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2099-01-03 (Estimated)

PRIMARY OUTCOMES:
Prospectively track patients who undergo cryoablation for breast cancer and record post-treatment related events. | five years from last participant enrollment
  record follow up of symptoms, reported complications, breast imaging findings, and results of any future biopsies related to cancer, and treatment of breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi S Kapoor, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States